CLINICAL TRIAL: NCT04786158
Title: Subcutaneous Apomorphine in the Treatment of Progressive Supranuclear Palsy and Cortico Basal Degeneration (APOPARKA)
Acronym: APOPARKA
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: CE_20200204_5_CHH
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Progressive Supranuclear Palsy; Corticobasal Degeneration
Keywords: pain; quality of life
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Corticobasal Degeneration; Pain | interventions — Apomorphine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Apomorphine — Reporting the effects of subcutaneous apomorphine on pain and on quality of life

SUMMARY:
Treatment of tauopathies such as Progressive Supranuclear Palsy (PSP) and Cortico Basal Degeneration (CBD) remains a major challenge. These rare severe neurodegenerative extrapyramidal movement disorders share phenotypic overlap and are usually painful. Parkinson disease (PD) is a common extrapyramidal movement disorder and continuous subcutaneous apomorphine infusion (CSAI) is commonly used in advanced PD patients to alleviate motor and non-motor fluctuations. Effects of subcutaneous apomorphine were investigated especially on pain and, on quality of life in 7 patients with PSD or CBD.This is an observational "real life" surveillance-based study.The Verbal Rating Scale for Pain (VRS) was used to assess changes in pain level and the clinical global impression-improvement scale (CGI-I) was used to assess changes in patient's illness before and during six months of treatment. Detailed report of the symptoms and side effects has been recorded by home nurses throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* PSP or CBD patients for whom a treatment with subcutaneaous apomorphine is indicated

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patient under a legal protection procedure
* Patient denying to participated to the study
* Lack of affiliation to a social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PSP or CBD patients for whom a treatment with subcutaneaous apomorphine is indicated
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Effects of subcutaneous apomorphine on pain | 6 months
  The Verbal Rating Scale for Pain (VRS) was used to assess changes in pain level. The VRS is a five-point scale and consists of a list of adjectives describing various levels of symptom intensity: 0= no itch, 1= mild itch, 2= moderate itch , 3= severe itch and 4=very severe itch. It is used to categorize the itch intensity and features high reliability and concurrent validity. VRS scale was assess before and during six months of treatment.
Effects of subcutaneous apomorphine on quality of life | 6 months
  The clinical global impression-improvement scale (CGI-I) was used to assess changes in patient's illness. The CGI-I is a 7 point scale that assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment." CGI-I scale was assess before and during six months of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Fondation Adolphe de Rothschild, Paris, Île-de-France Region, France